CLINICAL TRIAL: NCT01072461
Title: Optimizing Hand Rehabilitation Post-Stroke Using Interactive Virtual Environments
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Jersey Institute of Technology (Other)
Collaborators: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sergei V. Adamovich PhD, Associate Professor, New Jersey Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01HD058301-02 (NIH)
Record Dates: First submitted 2010-02-16; First posted 2010-02-22 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Cerebrovascular Accident; Hemiparesis; Hemiplegia
Keywords: Cerebrovascular Accident; Robotics; Virtual Reality; Rehabilitation; Neuroplasticity
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Train Paretic Hand and Arm Separate (Active Comparator): Eight three hour training sessions of robotically facilitated hand and arm training in complex virtual environments, using activities that train the fingers in isolation and other activities that train the arm in isolation.
  Interventions: Behavioral: HAS Training
- Train Paretic Hand and Arm Together (Experimental)
  Interventions: Behavioral: HAT training
- Train Both Hands Together in VE (Experimental)
  Interventions: Behavioral: Bimanual Training

INTERVENTIONS:
Behavioral: HAS Training — Robotically measured and facilitated training of the hemiparetic hand and arm in isolation, in a three dimensional haptically rendered virtual environment.
  Other Names: Isolated UE training
  Arms: Train Paretic Hand and Arm Separate
Behavioral: HAT training — Robotically measured and facilitated training of the hemiparetic hand and arm as an integrated functional unit, in a three dimensional haptically rendered virtual environment
  Other Names: Integrated UE training
  Arms: Train Paretic Hand and Arm Together
Behavioral: Bimanual Training — Robotically measured and facilitated training of the hemiparetic hand and non-hemiparetic hand together, in a three dimensional haptically rendered virtual environment
  Other Names: Bilateral UE training
  Arms: Train Both Hands Together in VE

SUMMARY:
The complexity of sensorimotor control required for hand function as well as the wide range of recovery of manipulative abilities makes rehabilitation of the hand most challenging. The investigators past work has shown that training in a virtual environment (VE) using repetitive, adaptive algorithms has the potential to be an effective rehabilitation medium to facilitate motor recovery of hand function. These findings are in accordance with current neuroscience literature in animals and motor control literature in humans. The investigators are now in a position to refine and optimize elements of the training paradigms to enhance neuroplasticity. The investigators first aim tests if and how competition among body parts for neural representations stifles functional gains from different types of training regimens. The second aim tests the functional benefits of unilateral versus bilateral training regimens.The third aim tests whether functional improvements gained from training in a virtual environment transfer to other (untrained) skills in the real world.

DETAILED DESCRIPTION:
The complexity of sensorimotor control required for hand function as well as the wide range of recovery of manipulative abilities makes rehabilitation of the hand most challenging. The investigators past work has shown that training in a virtual environment (VE) using repetitive, adaptive algorithms has the potential to be an effective rehabilitation medium to facilitate motor recovery of hand function. These findings are in accordance with current neuroscience literature in animals and motor control literature in humans. The investigators are now in a position to refine and optimize elements of the training paradigms to enhance neuroplasticity. The investigators first aim tests if and how competition among body parts for neural representations stifles functional gains from different types of training regimens. The second aim tests the functional benefits of unilateral versus bilateral training regimens.The third aim tests whether functional improvements gained from training in a virtual environment transfer to other (untrained) skills in the real world.

ELIGIBILITY:
Inclusion Criteria:

* Six months post cerebrovascular accident
* Residual upper extremity impairment that affects participation
* At least ten degrees of active finger extension
* Tolerate passive shoulder flexion to chest level

Exclusion Criteria:

* Severe neglect
* Severe aphasia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Jebsen Test of Hand Function | Two Weeks Prior to Training, Immediately Prior to Training, Immediately After Training, 3 Months After Training

SECONDARY OUTCOMES:
Change in Wolf Motor Function Test | Two Weeks Prior to Training, Immediately Prior to Training, Immediately After Training, 3 Months After Training
Change in 9 Hole Peg Test | Two Weeks Prior to Training, Immediately Prior to Training, Immediately After Training, 3 Months After Training
Change in Box and Blocks Test | Two Weeks Prior to Training, Immediately Prior to Training, Immediately After Training, 3 Months After Training
Change in Robotically Collected Kinematics | 1 day before training and 1 day after training
Change in Reach to Grasp Test | 1 day before training and 1 day after training

CONTACTS AND LOCATIONS:
Overall Officials: Sergei V. Adamovich, PhD, Principal Investigator — New Jersey Institute of Technology
Locations (1):
- New Jersey Institute of Technology, Newark, New Jersey, United States

REFERENCES:
- [Background] Adamovich SV, Fluet GG, Tunik E, Merians AS. Sensorimotor training in virtual reality: a review. NeuroRehabilitation. 2009;25(1):29-44. doi: 10.3233/NRE-2009-0497. PMID 19713617
- [Background] Tunik E, Adamovich SV. Remapping in the ipsilesional motor cortex after VR-based training: a pilot fMRI study. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:1139-42. doi: 10.1109/IEMBS.2009.5335392. PMID 19965144
- [Background] Fluet GG, Merians AS, Qiu Q, Lafond I, Saleh S, Ruano V, Delmonico AR, Adamovich SV. Robots integrated with virtual reality simulations for customized motor training in a person with upper extremity hemiparesis: a case study. J Neurol Phys Ther. 2012 Jun;36(2):79-86. doi: 10.1097/NPT.0b013e3182566f3f. PMID 22592063
- [Background] Tunik E, Saleh S, Adamovich SV. Visuomotor discordance during visually-guided hand movement in virtual reality modulates sensorimotor cortical activity in healthy and hemiparetic subjects. IEEE Trans Neural Syst Rehabil Eng. 2013 Mar;21(2):198-207. doi: 10.1109/TNSRE.2013.2238250. Epub 2013 Jan 9. PMID 23314780
- [Background] Bagce HF, Saleh S, Adamovich SV, Krakauer JW, Tunik E. Corticospinal excitability is enhanced after visuomotor adaptation and depends on learning rather than performance or error. J Neurophysiol. 2013 Feb;109(4):1097-106. doi: 10.1152/jn.00304.2012. Epub 2012 Nov 28. PMID 23197454
- [Background] Bagce HF, Saleh S, Adamovich SV, Tunik E. Visuomotor gain distortion alters online motor performance and enhances primary motor cortex excitability in patients with stroke. Neuromodulation. 2012 Jul;15(4):361-6. doi: 10.1111/j.1525-1403.2012.00467.x. Epub 2012 Jun 1. PMID 22672345
- [Background] Saleh S, Adamovich SV, Tunik E. Resting state functional connectivity and task-related effective connectivity changes after upper extremity rehabilitation: a pilot study. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:4559-62. doi: 10.1109/EMBC.2012.6346981. PMID 23366942
- [Background] Saleh S, Adamovich SV, Tunik E. Mirrored feedback in chronic stroke: recruitment and effective connectivity of ipsilesional sensorimotor networks. Neurorehabil Neural Repair. 2014 May;28(4):344-54. doi: 10.1177/1545968313513074. Epub 2013 Dec 26. PMID 24370569
- [Background] Yarossi M, Adamovich S, Tunik E. Sensorimotor cortex reorganization in subacute and chronic stroke: A neuronavigated TMS study. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:5788-91. doi: 10.1109/EMBC.2014.6944943. PMID 25571311
- [Background] Schettino LF, Adamovich SV, Bagce H, Yarossi M, Tunik E. Disruption of activity in the ventral premotor but not the anterior intraparietal area interferes with on-line correction to a haptic perturbation during grasping. J Neurosci. 2015 Feb 4;35(5):2112-7. doi: 10.1523/JNEUROSCI.3000-14.2015. PMID 25653367
- [Result] Qiu Q, Fluet GG, Lafond I, Merians AS, Adamovich SV. Coordination changes demonstrated by subjects with hemiparesis performing hand-arm training using the NJIT-RAVR robotically assisted virtual rehabilitation system. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:1143-6. doi: 10.1109/IEMBS.2009.5335384. PMID 19965145
- [Result] Adamovich SV, Fluet GG, Merians AS, Mathai A, Qiu Q. Incorporating haptic effects into three-dimensional virtual environments to train the hemiparetic upper extremity. IEEE Trans Neural Syst Rehabil Eng. 2009 Oct;17(5):512-20. doi: 10.1109/TNSRE.2009.2028830. Epub 2009 Aug 7. PMID 19666345
- [Result] Adamovich SV, Fluet GG, Mathai A, Qiu Q, Lewis J, Merians AS. Design of a complex virtual reality simulation to train finger motion for persons with hemiparesis: a proof of concept study. J Neuroeng Rehabil. 2009 Jul 17;6:28. doi: 10.1186/1743-0003-6-28. PMID 19615045
- [Result] Merians AS, Fluet GG, Qiu Q, Saleh S, Lafond I, Davidow A, Adamovich SV. Robotically facilitated virtual rehabilitation of arm transport integrated with finger movement in persons with hemiparesis. J Neuroeng Rehabil. 2011 May 16;8:27. doi: 10.1186/1743-0003-8-27. PMID 21575185
- [Result] Fluet GG, Merians AS, Qiu Q, Davidow A, Adamovich SV. Comparing integrated training of the hand and arm with isolated training of the same effectors in persons with stroke using haptically rendered virtual environments, a randomized clinical trial. J Neuroeng Rehabil. 2014 Aug 23;11:126. doi: 10.1186/1743-0003-11-126. PMID 25148846
- [Result] Fluet GG, Merians AS, Qiu Q, Rohafaza M, VanWingerden AM, Adamovich SV. Does training with traditionally presented and virtually simulated tasks elicit differing changes in object interaction kinematics in persons with upper extremity hemiparesis? Top Stroke Rehabil. 2015 Jun;22(3):176-84. doi: 10.1179/1074935714Z.0000000008. Epub 2015 Jan 22. PMID 26084322
- [Result] Puthenveettil S, Fluet G, Qiu Q, Adamovich S. Classification of hand preshaping in persons with stroke using Linear Discriminant Analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:4563-6. doi: 10.1109/EMBC.2012.6346982. PMID 23366943
- [Result] Boos A, Qiu Q, Fluet GG, Adamovich SV. Haptically facilitated bimanual training combined with augmented visual feedback in moderate to severe hemiplegia. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:3111-4. doi: 10.1109/IEMBS.2011.6090849. PMID 22254998
- [Result] Qiu Q, Adamovich S, Saleh S, Lafond I, Merians AS, Fluet GG. A comparison of motor adaptations to robotically facilitated upper extremity task practice demonstrated by children with cerebral palsy and adults with stroke. IEEE Int Conf Rehabil Robot. 2011;2011:5975431. doi: 10.1109/ICORR.2011.5975431. PMID 22275632
- [Result] Rohafza M, Fluet GG, Qiu Q, Adamovich S. Correlations between statistical models of robotically collected kinematics and clinical measures of upper extremity function. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:4120-3. doi: 10.1109/EMBC.2012.6346873. PMID 23366834
- [Result] Rohafza M, Fluet GG, Qiu Q, Adamovich S. Correlation of reaching and grasping kinematics and clinical measures of upper extremity function in persons with stroke related hemiplegia. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:3610-3. doi: 10.1109/EMBC.2014.6944404. PMID 25570772